CLINICAL TRIAL: NCT02867254
Title: Investigations of the Prevalence and Virulence of Candida Albicans in Periodontal and Endodontic Lesions in Diabetic and Normoglycemic Patients
Brief Title: Candida Albicans in Periodontal and Endodontic Lesions in Diabetic and Normoglycemic Patients
Acronym: diabetic
Status: Completed | Type: Observational
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Other Study IDs: Candida albicans
Record Dates: First submitted 2016-07-27; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes
Keywords: candida; endodontic lesion; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Torulopsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Groups1: 15 patients with type 2 diabetes mellitus with periodontal endodontic lesions
- Groups 2: 15 non-diabetics with periodontal endodontic lesions

SUMMARY:
Pulpal and periodontal tissues are closely related and have similar microbiota that cross-contamination between the pulp and periodontal tissues.The aim of this study was to investigate the prevalence of isolated Candida albicans from periodontal endodontic lesions in diabetic and normoglycemic patients and their virulence in different atmospheric conditions. A case-control study was conducted on 15 patients with type 2 diabetes mellitus (G1) and 15 non-diabetics (G2), with periodontal endodontic lesions. Samples of root canals and periodontal pockets were plated on CHROMagar for later identification by polymerase chain reaction (PCR) and virulence test.

DETAILED DESCRIPTION:
This case-control study was conducted on thirty patients (15 patients with type 2 diabetes mellitus and 15 normoglycemics) with clinical and radiographic diagnosis of a periodontal endodontic lesion. To assess the glycemic control of the patients were measured the plasma glucose level and glycosylated hemoglobin concentrations (HbA1c). All patients were initially submitted to examination to verify the clinical periodontal parameters (plaque index, probing bleeding, probing depth, clinical attachment level and gingival recession) and pulp sensitivity testing. The study included patients who presented periodontal pockets involving the apical region of the tooth and pulp necrosis (periodontal endodontic lesion). Exclusion criteria were: use of antibiotics in the last six months, pregnancy, smoking, other systemic diseases, clinical signs of oral candidiasis, and patients who did not sign a free and clarified consent term.

Sample collection Collection from the root canal was performed after access, rubber dam isolation, disinfection of the surgical field with 5.25% sodium hypochlorite, and neutralization with 5% sodium thiosulfato, with 3 sterile paper points remaining in the root canal for one minute. Sampling of the periodontal pocket was made at the deepest site through 3 sterile paper points, inserted one by one for one minute. The material collected from the periodontal pocket and the root canal was inoculated in Eppendorf tubes containing 1 ml of reduced transport fluid (RTF). Next, samples from each site were diluted and plated on the medium Saboraund Dextrose Agar plus Chloramphenicol and chromogenic medium (CHROMagar Candida ®, BioMerieux, Paris, France) and incubated at 37° C for 48h in a reduced oxygen atmosphere (10% CO2 and 90% air). The green colonies that grew on CHROMagar plates were chosen at random and stored in glycerol at 20° C for later identification by PCR.

ELIGIBILITY:
Inclusion Criteria:

-patients who presented periodontal pockets involving the apical region of the tooth and pulp necrosis (periodontal endodontic lesion).

Exclusion Criteria:

* use of antibiotics in the last six months,
* pregnancy,
* smoking,
* other systemic diseases,
* clinical signs of oral candidiasis
* patients who did not sign a free and clarified consent term.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim of this study was to investigate the prevalence of isolated Candida albicans from periodontal endodontic lesions in diabetic and normoglycemic patients and their virulence in different atmospheric conditional. A case-control study was conducted on 15 patients with type 2 diabetes mellitus (G1) and 15 non-diabetics (G2), with periodontal endodontic lesions. Samples of root canals and periodontal pockets were plated on CHROMagar for later identification by polymerase chain reaction (PCR) and virulence test.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sample collection from the root canal | 6 weeks
  Collection from the root canal was performed after access, rubber dam isolation, disinfection of the surgical field with 5.25% sodium hypochlorite, and neutralization with 5% sodium thiosulfato, with 3 sterile paper points remaining in the root canal for one minute.
Sample collection from the periodontal pocket | 6 weeks
  Sampling of the periodontal pocket was made at the deepest site through 3 sterile paper points, inserted one by one for one minute. The material collected from the periodontal pocket and the root canal was inoculated in Eppendorf tubes containing 1 ml of reduced transport fluid (RTF).

IPD SHARING:
Plan to Share IPD: Yes